CLINICAL TRIAL: NCT07235579
Title: Understanding Cauda Equina Syndrome:
Brief Title: Understanding Cauda Equina Syndrome
Acronym: UCES
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); University Hospitals of Derby and Burton NHS Foundation Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); East Kent Hospitals University NHS Foundation Trust (Other Government); Somerset NHS Foundation Trust (Other); Buckinghamshire Healthcare NHS Trust (Other); Milton Keynes University Hospital NHS Foundation Trust (Other Government); The Ipswich Hospital NHS Trust (Other); King's College Hospital NHS Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); Royal Devon and Exeter NHS Foundation Trust (Other); Royal Cornwall Hospitals Trust (Other); Walton Centre NHS Foundation Trust (Other); South Tees Hospitals NHS Foundation Trust (Other); Lancashire Teaching Hospitals NHS Foundation Trust (Other); City Hospitals Sunderland NHS Foundation Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government); The Leeds Teaching Hospitals NHS Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Nottingham University Hospitals NHS Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); North Bristol NHS Trust (Other); University Hospital Plymouth NHS Trust (Other); Barts & The London NHS Trust (Other); Barking, Havering and Redbridge University Hospitals NHS Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); University College London Hospitals (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 160318
Record Dates: First submitted 2019-05-08; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-06

CONDITIONS: Cauda Equina Syndrome
MeSH Terms: conditions — Cauda Equina Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cauda Equina Syndrome: For inclusion in this study, the patient must:
  * be over 18 years old;
  * be admitted to a specialist spinal service in the UK between 1st June 2018 and 31st May 2019;
  * have capacity to provide informed consent for participation in this study; and
  * have a diagnosis of clinical CES and structural compression of the cauda equina on imaging as determined by the treating clinician.
    * Clinical CES includes any disturbance of saddle sensation, bladder function, bowel function, sexual dysfunction and bilateral sciatica associated with radiological compression of the cauda equina. The cauda equina compression can be due to any cause, including, but not limited to, disc, tumour, infection, etc.

SUMMARY:
Cauda equina syndrome is a potentially devastating condition caused by compression of the cauda equina nerve roots. This can result in bowel, bladder and sexual dysfunction plus lower limb weakness, numbness, and pain. Cauda equina syndrome occurs infrequently but has serious potential morbidity and medico-legal consequences. This study aims to identify and describe the presentation and management of patients with cauda equina syndrome in the United Kingdom using trainee research collaborative networks. This will provide accurate incidence figures, establish current clinical practice, allow assessment of the adherence to national published standards of care, and determine patient outcomes from this condition. Accurate, up to date information about the presentation, management, and outcome of patients with cauda equina syndrome will inform standards of service design and delivery for this important but infrequent condition and help to identify future research priorities.

DETAILED DESCRIPTION:
Understanding Cauda Equina Syndrome (UCES) is a prospective cohort study of patients with confirmed CES managed at specialist spinal centres in the UK.

Cases will be identified by neurosurgical or orthopaedic trainees in each specialist centre through daily screening of tertiary referrals and admissions to specialist spinal services. All patients managed as CES by the treating team will be included in this audit. CES will be divided into CES suspected (CESS), CES incomplete (CESI), and CES retention (CESR).

Data regarding timing and type of symptom onset, referral, investigation, management, and outcome will be recorded anonymously on a secure database by the local trainee investigator during the patient's hospital admission and after discharge. Patient consent will be sought for the use of their data and patients will be asked to complete patient reported outcome measures representing their condition before surgery and up to one year after surgery. This data will be compared with care quality statements and published outcome data for CES.

The study will recruit for one year. Cases will be identified from admissions to spinal units between 1st June 2018 until 31st May 2019. The last one year follow up assessments will be sent to participants on 1st June 2020.

This is an observational study. No changes to routine patient care will occur during this study.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in this study, the patient must:

  * be over 18 years old;
  * be admitted to a specialist spinal service in the UK between 1st June 2018 and 31st May 2019;
  * have capacity to provide informed consent for participation in this study; and
  * have a diagnosis of clinical CES and structural compression of the cauda equina on imaging as determined by the treating clinician.

    * Clinical CES includes any disturbance of saddle sensation, bladder function, bowel function, sexual dysfunction and bilateral sciatica associated with radiological compression of the cauda equina. The cauda equina compression can be due to any cause, including, but not limited to, disc, tumour, infection, etc.

Exclusion Criteria:

* • Patients under 18 years old

  * Patients undergoing emergent decompression for unilateral motor or sensory symptoms (eg foot drop), without clinical evidence of CES
  * Patients referred with suspected CES where the diagnosis is not confirmed, for example:

    o Patients with the clinical symptoms and signs of CES without radiological evidence of cauda equina compression
  * Patients not admitted to participating spinal centres in the UK
  * Patients admitted to a participating spinal centre before 1st June 2018 or after 31st May 2019
  * Patients who are unable to provide informed consent for participation in this study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All neurosurgical and orthopaedic units managing patients with CES in the UK will be invited to participate. All patients admitted with radiologically confirmed CES will be identified by the lead local investigator via the screening of referral and admission systems at their spinal unit. All lead local investigators must be members of the clinical team caring for patients with CES in their unit.
  Capture-recapture methods will be used to ensure complete case ascertainment. In December 2018, June 2019, and December 2019 all local investigators will check their case ascertainment by asking their local coding departments for all discharges coded as CES using the diagnostic code ICD-10 G83.4.
Sampling Method: Non-Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
Identify the number of cases of Cauda Equina Syndrome (CES) in the UK in all collaborating centres | June 2018-June 2021
  Cases will be identified by neurosurgical or orthopaedic trainees in each specialist centre through daily screening of tertiary referrals and admissions to specialist spinal services. All patients managed as CES by the treating team will be counted.

SECONDARY OUTCOMES:
Describe the presenting symptoms and signs in patients with CES | June 2018-June 2021
  Study participants who have consented to participate will also be asked to fill out details about their patient journey to the spinal unit, their symptoms, patient reported outcome measures, and service usage. These will be collected electronically anonymously via the electronic database and linked to the patient record.
Describe the pathways of presentation to specialist spinal services for patients with CES in the UK and Ireland | June 2018-June 2021
  Patients will be asked about their care pathway prior to and after entering hospital
Describe the type and timing of investigation of patients with CES | June 2018-June 2021
  Timing of MRI scans will be gathered by a member of the local clinical care team. Time will be divided into hours from symptom onset (patient and clinician rated).
Describe the medical and surgical management of CES | June 2018- June 2021
  Type and timing of medical or surgical management of patients with cauda equina syndrome will be gathered by a member of the local clinical care team. Time will be divided into hours from symptom onset (patient and clinician rated), type will be a drop down menu of various types of operation and 'other' with room for explanation.
Describe clinical outcomes for patients with CES using validated patient reported outcome measures, stratified by presentation, investigations, and management | June 2018-June 2021
  Patient reported outcome measures will be used such as the ODI.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Woodfield, MBChB PhD, Study Chair — University of Edinburgh; Aimun Jamjoom, Study Director — University of Edinburgh; Ingrid Hoeritzauer, MBBChBAO, Study Director — University of Edinburgh
Locations (1):
- Department of Neurosciences, Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Ownership of the complete dataset arising from this study resides with the steering committee and the BNTRC. On completion of the study, the data will be analysed and tabulated, and a report will be prepared. Local data collected as part of this study belongs to the local team collecting that data.